CLINICAL TRIAL: NCT03947801
Title: Dairy Consumption During a High-intensity, High-volume Training Week in Young Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brock University (Other)
Responsible Party: Principal Investigator, PKlentrou, Professor and Associate Dean, Brock University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 18-289-Klentrou
Record Dates: First submitted 2019-05-08; First posted 2019-05-13 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Inflammatory Response; Sports Performance
Keywords: Greek Yogurt; Adolescent Athletes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Greek Yogurt condition (Experimental): 3x 160g of 0% Plain Greek yogurt (~115 kcals, 17 g protein, ~11.5 g carbs, 0 fat) consumed immediately following the training session, 1 h prior to bedtime, as well as one serving between breakfast and lunch on the subsequent day.
  Interventions: Other: Greek Yogurt
- Isoenergetic condition - Carbohydrate (Placebo Comparator): 3x 30g of isoenergetic CHO supplement (~115 kcal, 0.04 g protein, ~28.6 g carbs, 0 fat) consumed immediately following the training session, 1 h prior to bedtime, as well as one serving between breakfast and lunch on the subsequent day.
  Interventions: Other: Isoenergetic carbohydrate

INTERVENTIONS:
Other: Greek Yogurt — Female competitive soccer players (11-16y) will consume 0% plain Greek yogurt immediately following the training session, 1 h prior to bedtime, as well as one serving between breakfast and lunch on the subsequent day.
  Arms: Greek Yogurt condition
Other: Isoenergetic carbohydrate — Female competitive soccer players (11-16y) will consume an isoenergetic carbohydrate supplement immediately following the training session, 1 h prior to bedtime, as well as one serving between breakfast and lunch on the subsequent day.
  Arms: Isoenergetic condition - Carbohydrate

SUMMARY:
Our proposed study is a 5-d double-blind randomised cross-over trial, seeking to simulate a training identification camp in competitive adolescent soccer players

The purpose of the proposed study is to investigate whether increased protein consumption by Greek yogurt, compared to an isoenergetic carbohydrate (CHO) control supplement, consumed immediately following exercise training, prior to sleep and between breakfast and lunch, for a week during an intense training period (high volume, high intensity) will:

* Attenuate the pro-inflammatory response (cytokines, acute phase proteins)
* Reduced the severity of muscle damage and impairment (creatine kinase)
* Maintain performance

Secondary outcome measures:

- Increase bone turnover (in favour of formation)

DETAILED DESCRIPTION:
The proposed study is a randomized, double-blinded, cross-over trial. The protocol will consist of an information session, two identical training camps consisting of 5 consecutive days of intensified soccer training, differing only by nutritional intervention, and identical pre-and post-training session testing. Each testing block will be separated by 28-d to allow for an adequate wash-out and recovery period, during which participants would resume their regular soccer activities

Study Procedures:

All tests and measurements will be performed within eight-weeks. Specifically, participants will attend 1 information session, two identical pre- and post- training/testing sessions and two identical soccer specific training camps.

Information session:

One week prior to the initial soccer specific training camp, participants will be informed of all tests and procedures that will take place and be familiarized with all testing protocols.

Pre- and Post-training testing:

All participants will be tested twice: on the day before (pre) and day following (post) the 5-d soccer specific training camp. Specifically, Participants, will arrive at the University for pre- and post-training testing in the morning at the same time. Body composition measurements will be performed (e.g., standing/seated height, mass, % body fat) followed by fasted venous blood and saliva sampling. A standardized breakfast would then be provided followed by an adequate rest and digest period before performance testing (~1.5h). Performance testing would include a battery of soccer specific tests that cover, power (counter-movement jump, broad jump), speed (10m and 20m sprint), agility (modified 5-0-5) and aerobic capacity (beep-test). During both pre-and-post-testing sessions participants would consume the same standardised breakfast and perform the same tests in the same order for consistency amongst trials which would be repeated between the two testing blocks.

Soccer training:

The simulated 5-d soccer-specific training will be structured to mimic a heavy-volume, high-intensity training camp. Training sessions would occur at the same time each day in the evening for consistency. Drills/exercises will be administered by a certified technical soccer coach and knowledgeable training staff. Each session will began with a 15 min dynamic warm-up followed by 90 min of soccer-specific training, ending with a 15 min cool-down. The 90 min of soccer-specific training will be performed at maximal effort and consist of agility, sprinting and plyometric exercises as well as ball-handling, small-sided games (rondo) and shooting. Following each training session rating of perceived exertion (RPE) will be measured as an indicator of internal load.

Food/Drink supplement consumption:

During the study, three servings of 160 g of 0% plain GY (~115 kcals, 17 g protein, ~11.5 g carbs, 0 fat), or 30 g of isoenergetic CHO (~115 kcal, 0.04 g protein, ~28.6 g carbs, 0 fat) will be provided to participants immediately following the training session, 1 h prior to bedtime, as well as one serving between breakfast and lunch on the subsequent day. The yogurt will be sweetened or flavored with a non-caloric vanilla flavouring to match the taste of the control supplement. The CHO control supplement group will be an isoenergetic dose of a maltodextrin-based semi-solid pudding. This product will be made from non-fat vanilla pudding powder (1 part), maltodextrin (4 parts) and water. This product has been designed to resemble the consistency and texture of Greek yogurt.

Measurements

Questionnaires: Participant Screening and Medical History, Training History, Food frequency Questionnaire (FFQ), sessional RPE.

Anthropometric and body composition measurements: height, seated height, body mass and body fat percentage (%) using bioelectrical impedance analysis (BIA, InBody520; Biospace Co., Ltd., Seoul, S. Korea).

Somatic maturity: maturity offset (years from the age of peak height velocity) will be calculated based on height, seated height and weight measurements.

Exercise performance: will be examined prior to, as well as following each training intervention week. These tests are common in soccer and athletes are familiar with them. To limit confounding exercise influence on both biochemical and performance parameters, participants will be asked to refrain from other activities outside those prescribed to them during the training sessions and 48h prior to the initial pre-assessment visit.

Venous blood and saliva samples: will be collected on 4 separate occasions (24h prior and 24h following the last training session of each training intervention week). To control for circadian rhythm, the exercise session and related blood and saliva samples will be conducted at the same time of day. Saliva samples will be used to examine endocrine response. Venous blood samples will be used to examine inflammatory markers (cytokines - IL-6, IL-10 and TNF-α), c-reactive protein (CRP), IGF-I and indicators of muscle fatigue/damage (CK). Secondary measures may include irisin, oxidative stress (TBARS and ROS) and bone turnover by examining circulating markers of bone formation (PINP, Osteocalcin, BAP, OPG) and of bone resorption (CTX, TRAP, RANKL).

ELIGIBILITY:
Inclusion Criteria:

* Participant are female within the desired age ranges (11-16y)
* Participants are competitive soccer players
* Previous participation in high-performance training environment (periodization)

Exclusion Criteria:

* Participant is not female or falls outside of the desired age ranges (11-16y)
* Chronic/frequent use of medications that could affect inflammatory function - NSAIDS or Corticosteroids.
* Musculoskeletal injury - resulting in the inability to train and/or perform the baseline/post testing.

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Female adolescent competitive soccer players
Enrollment: 30 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-11-23 (Actual); Study Completion 2019-11-23 (Actual)

PRIMARY OUTCOMES:
Body mass (kg) | 8 weeks
  Anthropometric measures
Height (cm) | 8 weeks
  Anthropometric measures
Seated height (cm) | 8 weeks
  Used to calculate maturity offset in years from peak height velocity
Body fat (%) | 8 weeks
  Body composition
Rate of perceived exertion | 8 weeks
  1-10 scale of perceived exertion
Serum concentrations of BAP (ng/ml) | 8 weeks
  Bone formation marker
Serum concentrations of PINP (ng/ml) | 8 weeks
  Bone formation marker
Serum concentrations of OPG (pg/ml) | 8 weeks
  Bone formation marker
Serum concentrations of CTX (ng/ml) | 8 weeks
  Bone resorption marker
Serum concentrations of TRAP (ng/ml) | 8 weeks
  Bone resorption marker
Serum concentrations of RANKL (pg/ml) | 8 weeks
  Bone resorption marker
Plasma concentrations of irisin (ng/ml) | 8 weeks
  Plasma concentrations of pro-and-anti-inflammatory cytokines
Plasma concentrations of IL-6 (pg/ml) | 8 weeks
  Plasma concentrations of pro-and-anti-inflammatory cytokines
Plasma concentrations of IL-10 (pg/ml) | 8 weeks
  Plasma concentrations of pro-and-anti-inflammatory cytokines
Plasma concentrations of TNF-alpha (pg/ml) | 8 weeks
  Plasma concentrations of pro-and-anti-inflammatory cytokines
Plasma concentrations of CRP (pg/ml) | 8 weeks
  Plasma concentrations of pro-and-anti-inflammatory cytokines
Plasma concentration of creatine kinase (U/L) | 8 weeks
  Muscle damage

SECONDARY OUTCOMES:
Serum concentration of IGF-1 (pg/ml) | 8 weeks
  Serum concentration of IGF-1
Plasma concentration of TBARS | 8 weeks
  Oxidative stress
Plasma concentration of ROS | 8 weeks
  Oxidative stress
Saliva concentrations of cortisol (ug/dl) | 8 weeks
  Endocrine response
Saliva concentrations of testosterone (pg/ml) | 8 weeks
  Endocrine response
Oxidative stress | 8 weeks
  Plasma concentrations of markers of oxidative stress

OTHER OUTCOMES:
Aerobic Capacity - Beep Test | 8 weeks
  Aerobic capacity using the - Beep test; units - distance (m)
Maximal sprint ability | 8 weeks
  Maximal sprint ability using a 20 m sprint test; units - time (s)
Explosive leg power - Vertical jump performance | 8 weeks
  Explosive leg power using the counter-movement jump; units - height (cm)
Agility and Quickness | 8 weeks
  Agility using the 5-10-5 pro-agility test; units - time (s)

CONTACTS AND LOCATIONS:
Overall Officials: Panagiota Klentrou, PhD, Principal Investigator — Brock University
Locations (1):
- Elite soccer Development, Welland, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McKinlay BJ, Wallace PJ, Olansky S, Woods S, Kurgan N, Roy BD, Josse AR, Falk B, Klentrou P. Intensified training in adolescent female athletes: a crossover study of Greek yogurt effects on indices of recovery. J Int Soc Sports Nutr. 2022 Mar 22;19(1):17-33. doi: 10.1080/15502783.2022.2044732. eCollection 2022. PMID 35599913
- [Result] Klentrou P, McKee K, McKinlay BJ, Kurgan N, Roy BD, Falk B. Circulating Levels of Bone Markers after Short-Term Intense Training with Increased Dairy Consumption in Adolescent Female Athletes. Children (Basel). 2021 Oct 25;8(11):961. doi: 10.3390/children8110961. PMID 34828674